CLINICAL TRIAL: NCT04976400
Title: Research on Clinical Solutions of Artificial Joints for Men and Women With Different Designs and Semi-individual Total Knee Replacement：A Prospective Cohort Clinical Trial Study
Brief Title: Men and Women With Different Designs and Semi-individual Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Guizhou Orthopedics Hospital (Unknown); Shenyang Orthopedic Hospital (Other); West China Hospital (Other); Xi'an Honghui Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Jining Medical University (Other); Northern Jiangsu People's Hospital (Other); Inner Mongolia People's Hospital (Other); Shenzhen Pingle Orthopedics Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2021299
Record Dates: First submitted 2021-06-24; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-06

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Total knee replacement; gender
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Semi-individualized total knee arthroplasty
  Interventions: Procedure: semi-individualized total knee replacement treatment with a gender-specific design
- Control group (Active Comparator): Zimmer standard prosthesis total knee replacement
  Interventions: Procedure: Zimmer total knee replacement prostheses (Zimmer, Warsaw, IN, USA)

INTERVENTIONS:
Procedure: semi-individualized total knee replacement treatment with a gender-specific design — Patients in the experimental group received a semi-individualized total knee replacement treatment with a gender-specific design.
  Arms: test group
Procedure: Zimmer total knee replacement prostheses (Zimmer, Warsaw, IN, USA) — Patients in the control group received imported Zimmer total knee replacement prostheses (Zimmer, Warsaw, IN, USA).
  Arms: Control group

SUMMARY:
This study aims to evaluate the effectiveness of femoral condyle prosthesis, tibial tray prosthesis and meniscus prosthesis of semi-individualized total knee replacement prostheses designed with gender differences; and compare and analyze with the current classic prostheses, showing gender differences. The designed semi-personalized total knee replacement prosthesis lays the foundation for clinical application, including:

1. Compared with the classic osteotomy method, compare whether the semi-individualized total knee arthroplasty with a gender-specific design has advantages and better safety in the osteotomy method.
2. To evaluate the difference between the amount of osteotomy in the semi-individualized total knee arthroplasty designed for gender differences and the amount of classic osteotomy.
3. Compared with classic prostheses in the market, verify the clinical effects of semi-individualized total knee replacement prostheses designed for gender differences, and provide a basis for their clinical promotion and application.

DETAILED DESCRIPTION:
Patients meeting the inclusion and exclusion criteria were divided into the experimental group and the control group according to the patient's wishes. Patients in the experimental group received a semi-individualized total knee replacement treatment with a gender-specific design. The control group received imported Zimmer total knee replacement prostheses (Zimmer, Warsaw, IN, USA).

ELIGIBILITY:
Inclusion Criteria:

1. Various end-stage knee joint diseases such as degenerative osteoarthritis, traumatic arthritis or avascular necrosis, inflammatory joint disease, as well as correction of deformities, reconstruction after failure of some knee joint prostheses, and other techniques that cannot be handled In the case of fractures, total knee prosthesis replacement is required.
2. Age ≥50, ≤80 years old.
3. Subjects or guardians are willing and able to sign informed consent.

Exclusion Criteria:

1. History of previous knee surgery.
2. Severe knee deformity (valgus greater than 15° or valgus greater than 20°) or knee instability;
3. Severe flexion contracture deformity (flexion contracture> 25°);
4. Undertake total knee joint revision and replacement surgery;
5. Rheumatoid arthritis;
6. Body Mass Index (BMI)> 35.
7. Patients with neuromuscular insufficiency (such as paralysis, myolysis, or muscle weakness) can lead to postoperative knee instability or abnormal gait;
8. Pregnant or breastfeeding women;
9. Suffer from the underlying medical condition that the researcher believes that the patient is at an unacceptable risk (including but not limited to metabolism, hematology, kidney, liver, lung, nerve, endocrine, heart, infection, or gastrointestinal tract);
10. the current patient is not suitable Tests or severely progressive or uncontrolled diseases that put them at high risk, including any medical or psychiatric conditions that the investigator believes will prevent the subject from following the protocol or completing the study according to the protocol.
11. Being infected with human immunodeficiency virus (HIV), infectious hepatitis B or hepatitis C, or a corresponding medical history.
12. Suffering from a progressive infection or malignant disease, can provide chest X-ray, computed tomography (CT scan) or MRI evidence within 12 weeks before screening, and it is verified by a qualified physician.
13. Active systemic infections (except colds) or any other infections that will recur regularly during the previous two weeks.
14. A history of chronic or recurrent infectious diseases, or evidence of tuberculosis infection that was determined to be positive at the time of screening.
15. Subjects who have obtained positive or uncertain results can participate in the study if they have undergone a comprehensive tuberculosis examination (according to local practice/guidelines) within 12 weeks before baseline and finally confirmed that there is no evidence of active tuberculosis. If the presence of latent tuberculosis is confirmed, treatment must be initiated and maintained in accordance with local or national guidelines before the baseline.
16. History of lymphoproliferative disease, or any known malignancy, or history of malignancy of any organ system within the past 5 years (except for Bowen's disease, basal cell carcinoma, or actinic keratosis that has been treated and has no evidence of recurrence in the past 12 weeks ; Except for excised cervical carcinoma in situ or non-invasive malignant colon polyps).
17. Suffer from medical problems at the same time, including but not limited to the following: Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥95mmHg), congestive heart failure (New York Heart Association status classification III or IV).
18. Subjects with a serum creatinine level greater than 2.0 mg/dl (176.8 μmol/L). During screening, total white blood cell (WBC) count <2500/μL, or platelet <100000/μL or neutrophil <1500/μL or hemoglobin <8.5 g/dL.
19. During the six months before the baseline, there was a history of alcohol or drug abuse or evidence of ongoing abuse.
20. The patient is mentally incapable or unable to understand the requirements for participating in the research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
lower limb alignment | Before operation
  Full-length frontal radiographs of both lower extremities; both lower extremities and one-leg weight-bearing positive radiographs; （-3 3）is normal, The more out of this range, the worse.
lower limb alignment | 5 days after operation
  Full-length frontal radiographs of both lower extremities; both lower extremities and one-leg weight-bearing positive radiographs; （-3 3）is normal, The more out of this range, the worse.
lower limb alignment | 6 months after operation
  Full-length frontal radiographs of both lower extremities; both lower extremities and one-leg weight-bearing positive radiographs; （-3 3）is normal, The more out of this range, the worse.
lower limb alignment | 12 months after operation
  Full-length frontal radiographs of both lower extremities; both lower extremities and one-leg weight-bearing positive radiographs; （-3 3）is normal, The more out of this range, the worse.
Knee prosthesis position | 5 days after operation
  Coronal angle of femoral prosthesis and Coronal angle of tibial prosthesis，180° is normal. The more deviated from 180°, the worse.
Knee prosthesis position | 6 months after operation
  Coronal angle of femoral prosthesis and Coronal angle of tibial prosthesis，180° is normal. The more deviated from 180°, the worse.
Knee prosthesis position | 12 months after operation
  Coronal angle of femoral prosthesis and Coronal angle of tibial prosthesis，180° is normal. The more deviated from 180°, the worse.
Gait analysis | 5 days after operation
  Through the gait analysis platform and data acquisition system, Evaluate the patient's gait to achieve functional assessment of postoperative human movement.
Gait analysis | 6 months after operation
  Through the gait analysis platform and data acquisition system, Evaluate the patient's gait to achieve functional assessment of postoperative human movement.
Gait analysis | 12 months after operation
  Through the gait analysis platform and data acquisition system, Evaluate the patient's gait to achieve functional assessment of postoperative human movement.

SECONDARY OUTCOMES:
Operation time | during surgery
  from cutting the skin to completing the suture of the incision
The amount of bleeding | during surgery
  from cutting the skin to completing the suture of the incision
VAS score | Before operation
  Visual Analogue Scale/Score, the scale is 0-10 and 10 is worse.
VAS score | 5 days after operation
  Visual Analogue Scale/Score, the scale is 0-10 and 10 is worse.
VAS score | 6 months after operation
  Visual Analogue Scale/Score, the scale is 0-10 and 10 is worse.
VAS score | 12 months after operation
  Visual Analogue Scale/Score, the scale is 0-10 and 10 is worse.
KSS score | Before operation
  knee society score, the scale is 0-200 and 0 is worse.
KSS score | 5 days after operation
  knee society score, the scale is 0-200 and 0 is worse.
KSS score | 6 months after operation
  knee society score, the scale is 0-200 and 0 is worse.
KSS score | 12 months after operation
  knee society score, the scale is 0-200 and 0 is worse.
WOMAC score | Before operation
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, the scale is 0-100 and 100 is worse.
WOMAC score | 5 days after operation
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, the scale is 0-100 and 100 is worse.
WOMAC score | 6 months after operation
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, the scale is 0-100 and 100 is worse.
WOMAC score | 12 months after operation
  The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index, the scale is 0-100 and 100 is worse.
SF-36 score | Before operation
  short form 36 questionnaire, scale is 0-100 and 0 is worse.
SF-36 score | 5 days after operation
  short form 36 questionnaire, scale is 0-100 and 0 is worse.
SF-36 score | 6 months after operation
  short form 36 questionnaire, scale is 0-100 and 0 is worse.
SF-36 score | 12 months after operation
  short form 36 questionnaire, scale is 0-100 and 0 is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Jiakuo Yu, Doctor, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No